CLINICAL TRIAL: NCT00540215
Title: The Role of GLP-2 in Univercal Changes in Blood Flow in Humans
Brief Title: GLP-2 (Glucagonlike Peptide-2) and Blood Flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: H-D-2007-0050
Record Dates: First submitted 2007-10-04; First posted 2007-10-05 (Estimated); Last update posted 2011-02-11 (Estimated); Status verified 2007-10

CONDITIONS: Regional Blood Flow

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): 450 nmol GLP-2 SC
  Interventions: Other: Glucagonlike peptide
- 2 (Placebo Comparator): 1 ml isotonic saline SC
  Interventions: Other: Glucagonlike peptide

INTERVENTIONS:
Other: Glucagonlike peptide — 450 nmol native form, synthetic

SUMMARY:
It is the study aim to investigate the effect of glp-2 on blood flow in humans. we wish to study eventual changes in renal blood flow, carotic blood flow and cardiac out put.

GLP-2 will be administered subcutaneously, and the effect monitored by doppler ultra sound scannings and cotinuesly measuring of cardiac out put and blood pressure.

The study will include 15 healhty volunteers, 10 wil receive 450 nmol GLP-2 and 5 will receive 1 ml of isotonic saline (as baseline reference).

DETAILED DESCRIPTION:
se the above

ELIGIBILITY:
Inclusion Criteria:

* Age 20-60
* Healthy
* No medication
* Not pregnant

Exclusion Criteria:

* All of the persons not meeting the abowe mentioned criteria

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2007-10; Primary Completion 2008-01 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
effect of glp-2 | during study

SECONDARY OUTCOMES:
potential new ideas for further studies | months to years

CONTACTS AND LOCATIONS:
Overall Officials: lasse bremholm, MD, Principal Investigator — Glostrup university hospital
Locations (1):
- Glostrup University Hospital, Glostrup Municipality, Capital Region, Denmark